CLINICAL TRIAL: NCT06726213
Title: 'Walk and Talk - Connecting People With Psoriasis'. A Mixed-methods Exploratory Study to Determine Representativeness of Recruitment, Acceptability, and Feasibility of a Walk and Talk Intervention for People With Psoriasis
Brief Title: Walk and Talk: Connecting People With Psoriasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WALKANDTALK1.0
Record Dates: First submitted 2023-12-13; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Psoriasis; Social Isolation
MeSH Terms: conditions — Psoriasis; Social Isolation | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- walk and talk group (Experimental): Participants will participate in a walk and talk intervention once every two weeks for a 16-week period.
  Interventions: Other: Walk and talk
- Control group (No Intervention): Participants will continue their usual treatments.

INTERVENTIONS:
Other: Walk and talk — An hour long walk at a slow pace lead by a trained walking leader.
  Arms: walk and talk group

SUMMARY:
The main aim of this study is to determine the acceptability, representativeness (e.g. age, sex, ethnicity and body mass index) and ideal format of a Walk and Talk intervention for people with psoriasis.

Secondary aims are determining outcome measures of the intervention (patient related outcome measures, social connectedness, physical activity, cardiovascular risk)

Other objectives are to determine relevant outcome measures and sample size needed to statistically evaluate a future, larger study. There have been no similar studies evaluating social interventions in people with psoriasis, so an exploratory study is needed to calculate how many people are needed to participate. Measures will include social connectedness (loneliness), physical activity, cardiovascular risk, psychological wellbeing, quality of life and psoriasis severity.

Psoriasis is a systemic disease with multiple co-existent health issues. People with psoriasis are more socially isolated and inactive than the general population.

The health implications of social isolation are now recognised and thought to be equivalent to smoking. Consequently social prescribing is increasingly used for people living with long-term conditions. Specifically group walking activities are effective at increasing physical activity and improving mood. Additionally, disease specific walking groups provide peer psychosocial support.

It seems likely that a group walking intervention for people with psoriasis could promote social connectedness, increase physical activity and provide peer psychosocial support. However, as people with psoriasis avoid social contact, have low levels of physical activity and difficulty in discussing feelings, it is possible a Walk and Talk activity may not be taken up by many, or only by specific sub-groups such as young, slim, white people. Hence the need for an exploratory study before committing to a larger adequately powered study. Ultimately the investigators anticipate a format for Walk and Talk groups that is specifically tailored for people with psoriasis may enable groups to be rolled out at centres nationwide

DETAILED DESCRIPTION:
STUDY DESIGN 1. 'Walk and Talk - connecting people with psoriasis' is a mixed-methods exploratory study to determine the representativeness of recruitment, acceptability, and feasibility of a walk and talk intervention for people with psoriasis.

STUDY GROUP 2. Adult patients with a diagnosis of psoriasis +/- psoriatic arthritis attending the Dermatology Department at the Royal Free NHS Trust, London will be recruited for study. Participants must be able to walk for 1 hour at a slow pace (Can participants walk around 2km in an hour), or be a wheelchair user with someone who can push up hills if necessary (the study will not provide carers for wheelchair users, if a wheelchair user wishes to participate they must bring someone who is able to help them).

METHODS

1. RECRUITMENT In order to reduce bias and maximise inclusion, an 'opt-out' study design has been chosen. All patients who have attended the Royal Free London NHS Foundation Trust Psoriasis service within the last 2 years will be sent information about the study.

   * If a patient does not wish to participate, they will be able to opt-out of the study and will not be contacted again.
   * All patients who have not opted out will be invited to meet with an investigator to discuss entry into the study
   * If after 3 attempts to contact a patient regarding the study, no response is obtained, they will not be contacted again.
   * All individuals, who have not opted out, will be offered an appointment with a member of the research team. At this appointment there will be an opportunity for further discussion and questions about the study. The investigator will go through the information sheet with the potential participant.
   * Eligible and willing patients will be consented to participate in the study.

   Choosing not to participate will not alter their current or future care in any way.

   The 'opt out' study design has been chosen so the investigators can see if the people who participate in the study are representative of the overall population of patients who attend the Royal Free Hospital Psoriasis service. The investigators are keen to understand whether a social intervention such as a Walk and Talk intervention is acceptable to all subgroups of patients particularly with respect to ethnicity, gender, age and body mass index (weight).
2. INTERVENTION

   1. RANDOMISATION RANDOMISATION: Participants who have consented to participate in the study will be randomised using a computer-generated randomisation process to either a control group or a Walk and Talk (intervention) group at a 1:1 ratio.

      Participants who are in the intervention group will be allocated to a specific Walk and Talk group based on time and day of the week that is most convenient for them.

      A control group is included as this is an exploratory study. There have not been previous studies exploring the effect of a social intervention on people with psoriasis. The investigators are therefore interested to see potential areas for further investigation, such as improvement in quality of life, or social connectedness. The investigators need a control group to explore what differences there are for people participating in the social intervention, compared with those who are not participating in the intervention.
   2. BASELINE DATA COLLECTION (Time point 1) All participants will attend at a separate time to their usual dermatology outpatient appointment at the Royal Free Hospital to have baseline data collected (Time Point 1 - Figure 1). This will take approximately 30 mins. Questionnaires are validated questionnaires used in previous studies (Appendix 1.). Data collection will comprise of a variety of assessments to measure demographic, cardiovascular risk, disease severity quality of life, mood and wellbeing, lifestyle and medication.

Assessments for the control and the intervention groups will be at 4 time points:

1. Baseline
2. After 4 walk and talk sessions, (week 8) of the study; A short (15 minute) telephone interview will be performed for the participants in the intervention group to determine if any changes to the format of the Walk and Talk Intervention need to be made.
3. At completion of the 8 session Walk and Talk intervention (week 16 of study) Some participants in the intervention group will be randomly selected using the same randomisation process as described earlier to participate in an in-depth semi-structured interview). All participants will have the same data collected as they did in the baseline data collection.
4. 3 months after the end of the 8 session Walk and Talk intervention (week 28 of study), all participants will have their data collected again as they did in baseline, participants in the intervention group will out an additional questionnaire to assess whether they have continued to use the intervention after the end of the study.

Semi-structured interview:

Semi-structured digitally recorded interviews will be conducted by a member of the research team. Questions will focus on the participants' experience of the Walk and Talk intervention. Areas they enjoyed, changes they'd make for future interventions and any positive changes they've experiences as a result of the intervention. (see Appendix). The next round of 'Walk and Talk' interventions will be adapted according to feedback from these interviews.

INTERVENTION GROUP:

The intervention is a Group Walking Intervention (Walk and Talk Group), led by a trained walking leader who will be external to the trust. The walking leader will have no access to participant information other than a list of names of the participants in their particular group. The 'Walk and Talk' group will meet on 8 occasions for 1 hour to walk outside in a park every 2 weeks, it will take place on the same day/time and comprise of the same group participants and walk leader. There will be 8-10 participants in each group. It will involve walking with some simple stretches. The speed of the walk will be guided by the group level.

Each member of the intervention group will:

(i) Attend a virtual 'meet and greet' meeting with their group members (ii) Watch a short film about living with psoriasis at the end of the virtual meet and greet session (iii) Attend 8 x 1 hour outdoor walking sessions as above

Meet and Greet Zoom Call A week prior to the first Walk and Talk session, a Zoom 'meet and greet' call will be arranged where members of the group and the group leader will meet virtually for the first time. The session will be introduced by the PI who will be familiar to most participants and run by the study coordinator. Details of the study will be described briefly. Guidelines for behaviours and group responsibilities will be shared. Participants will be given the opportunity to ask questions. A psychologist will attend and silently observe.

Short Film Participants will be asked to watch the film 'Psoriasis: The Skin I'm In' at the end of the zoom call. The film is 11 minutes long and depicts true stories of people living with psoriasis. The aim of participants watching the film is to encourage discussion about psoriasis within the group. Focused groups suggested this be watched at home as it is quite emotional and would be difficult to watch in a group. The decision to ask participants to watch it as part of the zoom rather than completely independently is because it ensures a more focused environment and the investigators know that the film has been watched. To ensure participants feel comfortable, participants will be requested to turn off their cameras and microphones during the screening of the film. If they feel distressed they are able to leave the zoom without having to rejoin afterwards. A psychologist will be attending the zoom call and will be available for participants to speak to if needed.

Members of each walking group will be invited to join a WhatsApp Group (see Appendix) to enable participants to meet outside of the designated Walk and Talk intervention and to allow information about any group changes to be communicated. This will be voluntary. A member of the research team will also be part of the group to monitor for any inappropriate behaviours.

Group members will sign a 'Code of Conduct' (see Appendix) regarding use of What's App and conversations during the group activity.

CONTROL GROUP Participants in the control group will continue to receive standard psoriasis care delivered by the hospital but will not enter into a Walk and Talk group.

OTHER PARAMETERS In this pilot study the investigators will determine factors affecting recruitment and retention in the study. The investigators will determine if study participants are representative of the wider population of patients attending the Royal Free Psoriasis Service eg in sex, age, BMI and ethnicity. The investigators will determine if attendance of the Walk and Talk groups is dependent on external factors such as the weather, time of year or time of day, the exercise professional or mixed or same sex groups. Or if attendance is governed by patient factors such as age or sex. Similar factors for on-going adherence to increased activity and group relationships will be examined.

3. ANALYSIS

1. Qualitative analysis Semi-structured post-intervention interviews Randomly selected individuals who have completed the Walk and Talk intervention will be contacted and asked for an informal interview to discuss their experience of participating in a Walk and Talk group. The interviews will be semi-structured (similar questions will be asked at each interview, but there will be scope for conversation to naturally evolve too). The interviews will be recorded and transcribed.

   At least 2 researchers will analyse the transcripts independently and identify key recurring themes. The number of participants who are called for interview will depend upon 'saturation of themes'. Once no new information is being gathered from participants, themes will be considered saturated and no more interviews will take place.

   Information gathered from the interviews will be used to inform the ideal design of a Walk and Talk intervention for people with psoriasis. This design can then be used for a future fully powered definitive study.
2. Quantitative analysis

Statistical analysis will be descriptive only as there have been no previous studies to determine how many participants are needed in order to draw statistically significant results from the data.

The investigators will use the data gathered from this study to determine meaningful primary and secondary endpoints for a future study and also to calculate how many participants are needed for a future study to be statistically significant ie perform a power calculation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Diagnosed with psoriasis
* Currently attending psoriasis services in secondary care
* Must be able to walk for 30 minutes at a slow pace (approx 2km). Or be a wheelchair user with a carer who can push up hills if necessary

Exclusion Criteria:

* Participants who are not capable of understanding the information leaflet or consent form and thus are unable to give informed consent.
* Participants who do not understand verbal explanations or written information given in English will be excluded, as a number of questionnaires need to be completed. The translation service provided to the hospital is usually telephone operated.
* Participants not able to walk at a slow pace for 30 minutes will be excluded or wheelchair users who do not have a carer who can help to push up hills.
* Children will be excluded from study as this study involves making social interactions and contact with adults. This would not be appropriate, as child protection screens will not be performed on participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-07-07 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Participant satisfaction of a of a Walk and Talk intervention for people living with psoriasis. | 3 months
  Found by looking at feedback and comments of participants in thematic analysis of semi-structured interview.

SECONDARY OUTCOMES:
General Practice Physical Activity Questionnaire | 3 months
  A 4-level scale measuring how long the participant spends doing various types of physical activity. From none - 3 hours. A higher score shows higher levels of physical activity.
Psoriasis Area and Severity Index | 3 months
  A 4-level scale where participants rate different symptoms of psoriasis from 0 mild - 4 severe. A higher score reflects worse disease severity.
Dermatology Life Quality Index (DLQI) questionnaire | 3 months
  A 4-level scale with questions about the participants skin condition. Answers are on a scale from 'very much' to 'not at all'. A higher score indicates poorer quality of life.
Medication Adherence Questionnaire (MAQ) | 3 months
  A 2-level scale where participants answer Yes of No to questions concerning their medication. A higher score reflects lower adherence.
To understand the participants' experience of a weekly 'walk and talk' activity | 3 months
  Thematic analysis of semi-structured interviews.
Body mass index | 3 months
  Weight in kilograms divided by height in metres squared
Abdominal circumference | 3 months
  Measures in centimetres
Blood pressure | 3 months
  Systolic and diastolic blood pressure will be taken using a blood pressure cuff. It will be recorded as systolic pressure over the diastolic pressure in mm/Hg
Resting heart rate | 3 months
  Will be counted by a member of the research team
The Simplifies Psoriasis Index | 3 months
  This scale is in 3 parts. Part 1 provides a score from 0-50 of psoriasis severity, a higher score means it's more severe. Part 2 measures psychosocial impact, the participant marks their answer on a horizontal line from 0-10 with a higher score reflecting a higher psychosocial impact. Part 3 records how the Psoriasis has behaved and been treated in the past with a series of tick boxes. Scored are combines and a higher score reflects a larger impact.
Hospital Anxiety and Depression Score | 3 months
  A 4-level scale measuring participants agreement to statements about mood and feelings. A higher score reflects higher levels of anxiety and depression.
Penn State Worry questionnaire | 3 months
  A 4-level scale measuring participants frequency of worrying from 'Not at all typical' to 'Very typical of me'. A higher score reflects higher levels of worry
Cantril Ladder scale | 3 months
  A scale from 1-10. Participants select their position based on satisfaction with their life. A higher score reflects more satisfaction.
Insomnia severity index | 3 months
  A 5-level scale with questions about quality of sleep. A higher score reflects higher levels of insomnia.
Alcohol use disorders identification test; primary care | 3 months
  A 4-level scale rating the frequency and volume of alcohol intake. A higher score reflects higher chance of alcoholism.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Free, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No